CLINICAL TRIAL: NCT04063371
Title: Self-Administered Gerocognitive Examination (SAGE) for the Early Detection of Cognitive Impairment at Primary Care Provider Visits
Brief Title: SAGE for the Early Detection of Cognitive Impairment at Primary Care Provider Visits
Status: Completed | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Douglas Scharre, Professor-Clinical, Ohio State University
Other Study IDs: NEW-33307
Record Dates: First submitted 2019-08-19; First posted 2019-08-21 (Actual); Results first posted 2021-07-19 (Actual); Last update posted 2024-05-14 (Actual); Status verified 2024-05

CONDITIONS: Cognitive Impairment
MeSH Terms: conditions — Cognitive Dysfunction

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Control Group 1: At least one location will serve as the control office and will continue to conduct their visits including screening for cognitive impairment as they normally do using their usual method based on the primary care provider's normal practice.
- Intervention Group: At least one different location will serve as the intervention office where all the providers, as their standard of care, use a standardized method for screening for cognitive impairment consisting of using the SAGE or eSAGE test and having a conversation with an individual who knows the patient well (if possible) to ascertain if a significant change (based on primary care provider opinion) occurred in the patient's cognitive skills over the previous year.
  Interventions: Other: Self-Administered Gerocognitive Examination (SAGE) or Electronic Self-Administered Gerocognitive Examination (eSAGE); Other: Informant Conversation
- Control Group 2: Control group 2 consists of patients handled by the intervention office who did not complete the SAGE or eSAGE.

INTERVENTIONS:
Other: Self-Administered Gerocognitive Examination (SAGE) or Electronic Self-Administered Gerocognitive Examination (eSAGE) — The Self-Administered Gerocognitive Examination (SAGE) is a reliable and valid assessment that is used to detect MCI and early dementia. It is a pen and paper assessment that has 4 interchangeable versions. The digital version of SAGE (eSAGE; commercially known as BrainTest®) is made for tablet use, consists of the identical test questions as SAGE, and is strongly associated with the validated SAGE.
  Groups: Intervention Group
Other: Informant Conversation — If possible, the provider will have a conversation with an individual who knows the patient will to ascertain if a significant change (based on primary care provider opinion) occurred in the patient's cognitive skills over the previous year.
  Groups: Intervention Group

SUMMARY:
Thus far no large randomized trial has demonstrated a correlation between screening and improved outcomes. This would need to be done to gain widespread acceptance of screening and case finding programs. Early detection of cognitive impairment could potentially result in the appropriate treatment of reversible cognitive impairment conditions or earlier initiation of pharmacological interventions for the management of a variety of other dementia or Mild Cognitive Impairment (MCI) conditions. A screening approach that reduces the number of false positive screens would improve the comfort level of physicians and patients with cognitive screening programs.

The investigators propose to use the Self-Administered Gerocognitive Examination (SAGE) and the Electronic Self-Administered Gerocognitive Examination (eSAGE) to identify patients who score in the cognitive impairment range during an office visit with their primary care provider. Conversation with an individual who knows the patient well (if possible) will be performed to ascertain a significant change in the patient's cognitive skills over the previous year. The investigators wish to determine if screening for cognitive impairment in this way leads to new diagnoses and management outcomes compared to a group of primary care providers who use their current usual method in screening for cognitive impairment during office visits.

DETAILED DESCRIPTION:
The Ohio State University Wexner Medical Center has over 100 primary care providers who see patients at 14 offices in central Ohio. These providers routinely see geriatric patients and routinely conduct Annual Wellness Visits.

At least two primary care offices will be involved in this trial. At least one location will serve as the control office and will continue to conduct their visits including screening for cognitive impairment as they normally do using their usual method based on the primary care provider's normal practice. At least one different location will serve as the intervention office where all the providers, as their standard of care, use a standardized method for screening for cognitive impairment consisting of using the SAGE or eSAGE test and having a conversation with an individual who knows the patient well (if possible) to ascertain if a significant change (based on primary care provider opinion) occurred in the patient's cognitive skills over the previous year.

Chart reviews will be conducted on all of the patients who meet the inclusion/exclusion criteria for the trial using a 60 day window from the initial visit. The demographics, medical history and list of current medications will be reviewed. SAGE or eSAGE test results and the primary care provider's opinion of the informant information regarding the patient's cognitive change over the previous year will be obtained. Additionally, the charts will be reviewed for the number of referrals for further evaluation/management of potential cognitive impairment (including lab work, neuroimaging, neuropsychology testing, neurology/psychiatry, occupational therapy, physical therapy, speech therapy, counseling, respite care, legal assistance (DPOA or living will), day care, home health, social work, financial planning, and cognitive research), the initiation of pharmacological interventions for the management of cognitive impairment and the diagnosis of cognitive impairment. Charts will also be screened to assess the number of follow up visits that were scheduled after the office visit for follow up regarding cognitive issues. For the intervention office, chart reviews will be conducted on patients who complete the SAGE or eSAGE and on patients who do not complete the SAGE or eSAGE. Possible reasons for why patients would not complete the SAGE or eSAGE include: time constraints, patient noncompliance and provider oversight.

There will be 2 control groups. Control group 1 consists of primary care offices that did not use SAGE or eSAGE for any of their patients and Control group 2 consists of patients handled by the intervention office who did not complete the SAGE or eSAGE. Intervention group consists of patients handled by the intervention office who did complete the SAGE or eSAGE.

SAGE and eSAGE test scoring will be compared between the intervention office and the research site.

Upon completion of the trial, the providers from the intervention group will be requested to complete a questionnaire to evaluate the practicality and ease of use of the SAGE and eSAGE test.

ELIGIBILITY:
Inclusion Criteria:

* Adults 65-89 years of age who complete a non-acute care office visit.

Exclusion Criteria:

* Diagnosis of mild cognitive impairment or dementia in the medical records.
* Diagnosis of visual loss or conditions causing visual loss in the medical records unless it is clear that the loss would not be sufficient to preclude reading standard medical forms with or without the use of visual aids.

Ages: 65 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: Adults 65-89 without a known diagnosis of cognitive impairment or dementia who complete a non-acute care office visit will be included in the trial.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Actual)
Dates: Start 2019-10-14 (Actual); Primary Completion 2020-04-06 (Actual); Study Completion 2020-07-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Douglas Scharre, MD, Principal Investigator — Ohio State University
Locations (1):
- The Ohio State University, Columbus, Ohio, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Scharre DW, Vrettos NE, Nagaraja HN, Wexler RK, Clark AD, Nguyen CM. Self-administered gerocognitive examination (SAGE) aids early detection of cognitive impairment at primary care provider visits. Front Med (Lausanne). 2024 Jun 13;11:1353104. doi: 10.3389/fmed.2024.1353104. eCollection 2024. PMID 38938387

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control Group 1 | Intervention Group | Control Group 2
Started | 100 | 100 | 100
Completed | 100 | 100 | 100
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control Group 1 | Intervention Group | Control Group 2 | Total
Number analyzed (Participants) | 100 | 100 | 100 | 300
Age, Continuous [Median (Full Range); unit: years] | 70.0781 [65.03898 to 89.63086] | 71.46759 [65.02529 to 87.30375] | 71.53598 [65.03613 to 88.75462] | 70.88031 [65.02529 to 89.63086]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 57 | 58 | 67 | 182
  Male | 43 | 42 | 33 | 118
Race/Ethnicity, Customized [Number; unit: participants]
  African American | 10 | 16 | 22 | 48
  Caucasian | 82 | 83 | 74 | 239
  Other | 8 | 1 | 4 | 13
Region of Enrollment [Number; unit: participants]
  United States | 100 | 100 | 100 | 300

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With a Diagnosis of a Cognitive Impairment Disorder Measured by Pharmacological Interventions for the Management of Cognitive Impairment.
Description: Number of participants in the intervention and the two control groups with diagnosis of a cognitive impairment disorder as measured by pharmacological interventions for the management of cognitive impairment.
Time Frame: 60 days
Measure: Number; unit: participants
Arm/Group | Control Group 1 | Intervention Group | Control Group 2
Number analyzed (Participants) | 100 | 100 | 100
participants | 0 | 0 | 0

2. Primary Outcome: Number of Participants in the Intervention and Control Groups With Any Referral for Further Evaluation/Management of Potential Cognitive Impairment
Description: Number of participants in the intervention and the two control groups with any referral for further evaluation/management of potential cognitive impairment.
Time Frame: 60 days
Measure: Number; unit: participants
Arm/Group | Control Group 1 | Intervention Group | Control Group 2
Number analyzed (Participants) | 100 | 100 | 100
participants | 2 | 7 | 0

3. Primary Outcome: Number of Participants in the Intervention and the Control Groups With at Least One Follow-up Visit for Additional Investigation of a Cognitive Impairment Disorder.
Description: Number of participants in the intervention and the two control groups with at least one follow-up visit for additional investigation of a cognitive impairment disorder.
Time Frame: 60 days
Measure: Number; unit: participants
Arm/Group | Control Group 1 | Intervention Group | Control Group 2
Number analyzed (Participants) | 100 | 100 | 100
participants | 1 | 4 | 0

4. Secondary Outcome: Number of Referrals Used for Subjects in the Intervention and Control Groups for Further Evaluation/Management of Potential Cognitive Impairment.
Description: Number of referrals used for subjects in the intervention and two control groups for further evaluation/management of potential cognitive impairment.
Time Frame: 60 days
Population: The referrals that were investigated are listed in the rows below.100 subjects were analyzed in each group, but primary outcome measure 2 lists the total number of subjects in each group that had referrals. This secondary outcome measure lists the breakdown of the referrals. Some subjects had multiple referrals.
Measure: Number; unit: participants
Arm/Group | Control Group 1 | Intervention Group | Control Group 2
Number analyzed (Participants) | 100 | 100 | 100
participants
  Lab work | 1 | 2 | 0
  Neuroimaging | 1 | 4 | 0
  neuropsychological testing | 0 | 0 | 0
  neurology/psychiatry | 2 | 4 | 0
  occupational therapy | 0 | 0 | 0
  physical therapy | 0 | 0 | 0
  speech therapy | 0 | 0 | 0
  counseling | 0 | 3 | 0
  respite care | 0 | 0 | 0
  legal assistance | 0 | 2 | 0
  day care | 0 | 0 | 0
  home health | 0 | 2 | 0
  social work | 0 | 1 | 0
  financial planning | 0 | 1 | 0
  cognitive research | 0 | 0 | 0
  other | 1 | 6 | 0

5. Secondary Outcome: Number of Participants With Pharmacological Interventions for the Management of the Cognitive Impairment in the Subgroups of the Intervention Arm With and Without Additional Inputs From Informants
Description: Number of participants with pharmacological interventions for the management of the cognitive impairment in the two subgroups of the intervention arm with and without additional inputs from informants
Time Frame: 60 days
Population: Since no participants were started on pharmacological interventions for the management of cognitive impairment (results of primary outcome measure 1) this outcome measure was not applicable. No data was analyzed since the subgroup in question did not exist. 100 subjects in each group were analyzed for primary outcome measure #1. This secondary outcome measure was intended to further analyze the subgroup. 0 is entered for these results since the subgroup did not exist.
Arm/Group | Control Group 1 | Intervention Group | Control Group 2
Number analyzed (Participants) | 0 | 0 | 0

6. Secondary Outcome: Scoring
Description: Differences of SAGE and eSAGE scoring between intervention office and research site.
Time Frame: 60 days
Population: Only the SAGE was utilized in this trial. eSAGE was not utilized. 93 SAGEs were graded by the providers. The others were completed and were reviewed by the provider but did not have the provider's score documented. The researchers re-graded the 93 SAGEs and documented scoring discrepancies between the 2 offices. The included results represent the total score difference between the research office and the provider. The SAGE is scored from 0-22 with 0 being the lowest score.
Measure: Number; unit: SAGEs
Units Other Than Participants: SAGE tests
Arm/Group | Intervention Group
Number analyzed (Participants) | 93
Number analyzed (SAGE tests) | 93
SAGEs
  -7 score difference | 1
  -5 score difference | 1
  -4 score difference | 7
  -3 score difference | 13
  -2 score difference | 22
  -1 score difference | 25
  0 score difference | 19
  +1 score difference | 3
  +3 score difference | 2

7. Secondary Outcome: Questionnaires
Description: Results of the questionnaire to evaluate the practicality and ease of use of the SAGE and eSAGE test by primary care providers and staff.
Time Frame: 60 days
Measure: Count of Participants; unit: Participants
Groups:
- Providers: The providers from the intervention group were asked to complete a questionnaire to evaluate the practicality and ease of use of the SAGE and eSAGE test.
Arm/Group | Providers
Number analyzed (Participants) | 7
Participants
  Would recommend the SAGE test during office visits for other colleagues | 6
  Would not recommend the SAGE test during office visits for other colleagues | 1

ADVERSE EVENTS:
Time Frame: Adverse event collection was not applicable for this trial since it was a retrospective chart review study that compared standard of care practices. Although there was an intervention (SAGE or eSAGE) the intervention was a standard of care practice for one of the buildings. It was already in place by that office when we started our trial and was not implemented for the trial. We reviewed the charts retrospectively and compared standard of care practices.
Description: Adverse event collection was not applicable for this trial since it was a retrospective chart review study that compared standard of care practices. Although there was an intervention (SAGE or eSAGE) the intervention was a standard of care practice for one of the buildings. It was already in place by that office when we started our trial and was not implemented for the trial. We reviewed the charts retrospectively and compared standard of care practices. AE's were not monitored and were n/a.
Arm/Group | Control Group 1 | Intervention Group | Control Group 2
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-02-18): https://cdn.clinicaltrials.gov/large-docs/71/NCT04063371/Prot_SAP_000.pdf